CLINICAL TRIAL: NCT07304271
Title: Randomised Phase III Trial of First Line Intraperitoneal Paclitaxel and Systemic Therapy Versus Systemic Therapy Alone in Gastric Cancer Patients With Peritoneal Metastases - IPa-Gastric
Brief Title: Intraperitoneal Paclitaxel and Systemic Therapy Versus Systemic Therapy Alone in Gastric Cancer Patients With Peritoneal Metastasis
Acronym: IPa-Gastric
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Magnus Nilsson (Other)
Responsible Party: Sponsor-Investigator, Magnus Nilsson, Head of the Division of Surgery and Oncology, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-514879-17-00
Record Dates: First submitted 2025-11-19; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer Peritoneal Metastases
Keywords: Gastric cancer; Peritoneal metastasis; Intraperitoneal administration
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard systemic therapy (Active Comparator): The control arm treatment in the study will consist of standard investigator's choice therapy with systemic chemotherapy and any targeted therapies indicated in the standard clinical practice setting
  Interventions: Drug: Standard systemic therapy
- Intraperitoneal paclitaxel + Standard systemic therapy (Experimental): The experimental arm treatment will consist of the same standard systemic investigator's choice treatment described above combined with IP paclitaxel.
  Interventions: Drug: Intraperitoneal Paclitaxel; Drug: Standard systemic therapy

INTERVENTIONS:
Drug: Intraperitoneal Paclitaxel — Intraperitoneally administered Paclitaxel
  Arms: Intraperitoneal paclitaxel + Standard systemic therapy
Drug: Standard systemic therapy — Standard investigator's choice therapy with systemic chemotherapy and any targeted therapies indicated in the standard clinical practice setting

SUMMARY:
The most common site for gastric cancer distant metastases is the peritoneum. Median survival for this group of patients is short and systemic cytotoxic treatment response is poor, partly due to the low uptake of the treatment compounds to the peritoneum during systemic chemotherapy. Infusion of cytotoxic drugs directly into the abdominal cavity has been shown to have a high objective response rate and low toxicity. The IPa-Gastric trial is an open-label, multicentre, randomised, phase-III study in the first line setting in gastric cancer patients with peritoneal metastases. Patients will receive the study treatments until disease progression, unacceptable side effects, the investigator's decision to end treatment for other reasons, death, or end of study. After discontinuing study treatments, each patient will be followed up for all study endpoints that are clinically feasible, until death or end of study. The primary objective is to compare overall survival (OS) for patients randomised to intraperitoneal (IP) paclitaxel and standard ST versus those randomised to standard ST only.

ELIGIBILITY:
Inclusion Criteria:

* Gastric or gastro-oesophageal junction Siewert type II or III adenocarcinoma verified by biopsy or cytology from the primary tumour
* Peritoneal metastasis verified by biopsy, or cytology from ascites or peritoneal wash fluid
* Staging laparoscopy with assessment of peritoneal cancer index (PCI) performed less than four weeks before enrolment.
* Patients with tumour positive cytology (CYT+) without clinically manifest peritoneal metastases at baseline (PCI 0) staging laparoscopy can be included if they persist to be CYT+ after at least four cycles of systemic chemotherapy.
* Adequate hematology assessment and serum chemistry
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Age of at least 18 years
* Life expectancy of at least three months
* Assurance that adequate anti-reproductive measures will be taken during study interventions when applicable

Exclusion Criteria:

* Comorbidity that does not allow treatment with ST or IP paclitaxel
* Confirmed or suspected severe abdominal adhesions
* Severe coagulation disorder which precludes surgical interventions
* Distant metastases (including M1 lymph node metastases) other than peritoneal, with the specific exception of ovarian metastases
* Symptomatic ascites already requiring drainage for palliation, or expected to require drainage in the short term
* Peritoneal recurrence of gastric cancer diagnosed within 6 months after curative intent surgery
* Previously received more than 2 cycles of palliative-intent systemic chemotherapy (with the specific exception of cytology positive patients without manifest peritoneal metastases) for the current gastric cancer (up to 2 cycles of first line chemotherapy is allowed). Perioperative chemotherapy within previous curative context is allowed
* Another malignancy that can affect survival within the next three years
* Known or suspected allergies against any product included in the trial interventions
* DYPD deficiency
* Pregnancy or recent delivery within 28 days postpartum or ongoing breastfeeding
* Active sex-life without use of secure contraceptive method.
* If the investigator considers the patient inappropriate for participation in the study for any other reason
* Ongoing or recent participation (within 30 days) in a clinical trial with an investigational medicinal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Assessed every second month from randomization until study completion, during a maximum of 60 months.
  Overall survival (OS), defined as time from randomisation to death from any cause. For subjects who are still alive at the End of Study (EoS), or who are lost to follow up, OS time will be censored at the last recorded date that the subject was known to be alive.

SECONDARY OUTCOMES:
Treatment-related toxicity | Assessed continously from start of treatment until 4 weeks after end of treatment for respective participant, during a maximum of 61 months.
  Incidence of Adverse Events (AE) as assessed by CTCAE v5.0
General Health Related Quality of Life (HR QoL) | Assessed at baseline and 2, 4, 6, 12 and 24 months after randomisation
  General Health Related Quality of Life (HR QoL) as measured by the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire QLQ-C30. Two types of scores will be calculated: raw scores and linearly transformed scores.
Progression free survival (PFS) | Assessed from randomization until study completion, during a maximum of 60 months.
  PFS is defined as time from randomisation to first documentation of progression according to RECIST1.1, progression of peritoneal carcinomatosis index (PCI), radiological progression of ascites, need for drainage of ascites or death, whichever occurs first.
Radiological response of treatment on ascites present at baseline. | Assessed from baseline visit until study completion, during a maximum of 60 months.
  Observed and change from baseline values will be summarized descriptively at planned visits by treatment. A mixed-effects model repeated measures (MMRM) analysis will evaluate longitudinal change from baseline. The baseline score will be included as a covariate.
Paracentesis of ascites | Assessed from randomization until study completion, during a maximum of 60 months.
  Time from randomisation to first paracentesis of ascites
Amount of ascites drained | Assessed from time of randomisation to study completion, during a maximum of 60 months.
  The sum of the volume drained from each patient from the date of randomisation to date of death, censoring or end of study
Proportion of patients fulfilling the criteria for curative intent conversion surgery. | Assessed from randomisation until study completion, during a maximum of 60 months.
  Criteria for conversion surgery are 1. CYT- at two consecutive sampling occasions, 2. No signs of progression on radiology, 3. No macroscopic peritoneal disease visible at new staging laparoscopy, 4. Discussion at MDT with conversion surgery considered feasible.
The proportion of patients undergoing conversion surgery | Assessed from randomisation until study completion, during a maximum of 60 months.
  The proportion of patients actually undergoing conversion surgery

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Nilsson, MD, Professor, Study Director — Karolinska University Hospital
Locations (5):
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided
A plan for IPD sharing will be added later